CLINICAL TRIAL: NCT02037568
Title: Improved Behavioral Outcome in Allogeneic Hematopoietic Stem Cell Transplant Patients by Reducing Caregiver Distress: Behavioral and Physiological Evidence
Brief Title: Improved Outcome in Allogeneic Hematopoietic Stem Cell Transplant (HSCT) Patients by Reducing Caregiver Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2639
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Hematopoietic/Lymphoid Cancer
Keywords: depression; stress; caregiving; anxiety; psychoeducation intervention; psycho-oncology; allogeneic hematopoietic stem cell transplant
MeSH Terms: conditions — Hematologic Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caregiver Self-Directed (No Intervention): Orientation class; laboratory biomarker analysis; questionnaire administration; survey administration; treatment as usual psychosocial care; caregiver workbook.
- Caregiver Intervention (Experimental): Orientation class; laboratory biomarker analysis; questionnaire administration; survey administration; Psychoeducation and Relaxation (fPER), which included one-on-one psychoeducation, and stress management intervention.
  Interventions: Behavioral: fPER

INTERVENTIONS:
Behavioral: fPER — Briefly in order, the sessions will include: 1) Overview and introduction to stress management, 2) Stress and the mind-body connection, 3) How our thoughts can lead to stress, 4) Coping with stress, 5) Strategies for maintaining energy and stamina, 6) Coping with uncertainty and fear of unknown, 7) Managing changing relationships/communicating needs, and 8) Getting the support they need, modeled after a successful intervention for patient groups. Manualization is crucial for successful wider implementation. Sessions 9 and 10 will provide booster sessions in which the interventionist will assess current challenges for the caregiver, provide review, and emphasize further coping skills training that might assist the caregiver in managing current stressors such as coping with the "new normal."
  Other Names: Other Names:; "fone" PsychoEducation and Relaxation
  Arms: Caregiver Intervention

SUMMARY:
PURPOSE: As this is a randomized controlled trial, all subjects receiving stress management psychoeducation will be expected to obtain a new set of coping skills that will allow them to better deal with the stressors of caregiving for an allogeneic HSCT patient. It is expected that improving caregiver status will improve patient quality of life.

DETAILED DESCRIPTION:
Specific Aims

* Create a Community Advisory Board (CAB) consisting of allogeneic HSCT patients, caregivers, blood cancer oncologists, support staff and study investigators to provide input.
* Assess patient Quality of Life (QOL) following an allogeneic HSCT using the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) as the primary patient outcome. Patients whose caregivers receive "fone" PsychoEducation and Relaxation (fPER) will have improved QOL compared to caregivers assigned to treatment as usual (TAU).
* Test the impact of fPER on a caregiver composite distress score (encompasses depression, anxiety, and stress) as the primary caregiver outcome. Caregivers receiving fPER will have reduced distress.
* Assess biomarkers of allostatic load in patients prior to transplant and caregivers during the transplant process using novel biomarkers (hair cortisol and telomeres). fPER will be associated with reduced allostatic load in caregivers compared to TAU. Patient hair cortisol collected only before transplant will relate to QOL at intake.

OUTLINE: Caregivers are randomized to 1 of 2 groups.

All patients and caregivers, regardless of randomization, are informed of what to expect during the transplant process and how to locate available support resources within each program. Patients and caregivers are given information that is specific to their involvement in the transplantation process and recovery phase.

* Group I (treatment as usual [TAU]): Subjects randomized to TAU will be encouraged to participate in available support programs at their respective centers which are very similar between sites and include individual counseling as well as support groups. Due to the impact of our prior intervention on caregiver distress, we will provide each caregiver randomized to TAU a workbook prepared for someone to use without inclusion of one-on-one sessions with a therapist.
* Group II (PsychoEducation and Relaxation [fPER]): Caregivers will participate in the fPER intervention prior to transplant. The fPER consists of 10 sessions to include 4 weekly 60-minute sessions followed by 4 biweekly 60-minute sessions and two additional sessions between day 100 and 6 months post-transplant. Each fPER session will be devoted to a separate topic with the goal of assisting the caregiver in the development and application of stress-management coping skills including learning problem-solving skills, identifying cognitive distortions, application of relaxation techniques, use of the emWave2, coping skills training, effective use of social support, and establishing appropriate goals. All caregivers in fPER will be provided a Caregiver Workbook that includes information about the session topics and homework assignments. fPER sessions will be delivered either at the clinic during patient visits or via video chat. fPER will also include incorporation of Smartphone technology to make the interventionist available by video chat.

Caregivers and patients undergo psychosocial assessments prior to randomization, and at 6 weeks, 3 months and 6 months after transplant (anchored to the day of transplant as day 0). At each phase, patients and caregivers will complete the same battery of questionnaires that includes the Center for Epidemiological Studies-Depression scale (CES-D), the perceived stress scale (PSS), and the State-Trait Anxiety Inventory (STAI). Additionally the patient will complete the FACT-BMT each time while the caregiver completes the Caregiver Reaction Assessment (CRA) and Carer Support Needs Assessment Tool (CSNAT). The patient and the caregiver will additionally complete a demographic questionnaire that includes questions regarding age, diagnosis, income, and other standard questions regarding nutrition, health behaviors, and health services utilization. At study completion, an exit questionnaire will address each subject's evaluation of the study and the group in which they were assigned.

Blood and hair samples from caregivers will be collected every three months: baseline (patient and caregiver), 3 (caregiver) and 6 (patient and caregiver) months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* DISEASE CHARACTERISTICS (Meets all of the following criteria):

  * Patient undergoing allogeneic hematopoietic stem cell transplant (HSCT)
  * Caregiver: the person in the patient's life who is primarily responsible for care decisions, emotionally invested in the patient's care, provides instrumental care such as transportation, and available if randomized to the fPER group to participate in the majority of intervention sessions
* PATIENT CHARACTERISTICS:

  * Able to read and speak English
  * Has telephone access
* CAREGIVER CHARACTERISTICS:

  * Able to read and speak English
  * Willingness to use a Smartphone
  * No serious medical condition likely to influence cortisol assessment in their hair
  * Alcohol consumption limited to < 2 drinks/day
  * At least 18 years of age

Exclusion Criteria:

* PRIOR CONCURRENT THERAPY:

  * No history of a psychiatric illness unrelated to the HSCT within the past 18 months
  * No steroid medications (caregiver)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-01; Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Laudenslager, PhD, Principal Investigator — University of Colorado Denver (Anschutz Medical Campus)
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Presbyterian/St. Luke's Medical Center (PSLMC), Denver, Colorado

REFERENCES:
- [Derived] Sannes TS, Ranby KW, Yusufov M, Brewer BW, Jacobs JM, Callan S, Ulrich GR, Pensak NA, Natvig C, Laudenslager ML. More often than not, we're in sync: patient and caregiver well-being over time in stem cell transplantation. Health Qual Life Outcomes. 2022 Jan 10;20(1):6. doi: 10.1186/s12955-021-01909-3. PMID 35012566
- [Derived] Laudenslager ML, Simoneau TL, Mikulich-Gilbertson SK, Natvig C, Brewer BW, Sannes TS, Kilbourn K, Gutman J, McSweeney P. A randomized control trial of stress management for caregivers of stem cell transplant patients: Effect on patient quality of life and caregiver distress. Psychooncology. 2019 Aug;28(8):1614-1623. doi: 10.1002/pon.5126. Epub 2019 May 25. PMID 31127974

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregivers and their Allo-HSCT patients were recruited consecutively between 3/2014 and 11/2016 during pre-transplant screening admitted for treatment to two transplant programs in the Denver metro area for participation in this study: a university-based NCI-designated Comprehensive Cancer Center and a community-based cancer center.
Pre-assignment Details: 159 patient-caregiver dyads were consented (318 participants).
Groups:
- Caregiver Self-Directed (TAU): Orientation class; laboratory biomarker analysis; questionnaire administration; survey administration; treatment as usual psychosocial care; caregiver workbook.
- Caregiver Intervention (PEPRR 2.0): Orientation class; laboratory biomarker analysis; questionnaire administration; survey administration; Psychoeducation and Relaxation (fPER), which included one-on-one psychoeducation, and stress management intervention.
  fPER: Briefly in order, the sessions will include: 1) Overview and introduction to stress management, 2) Stress and the mind-body connection, 3) How our thoughts can lead to stress, 4) Coping with stress, 5) Strategies for maintaining energy and stamina, 6) Coping with uncertainty and fear of unknown, 7) Managing changing relationships/communicating needs, and 8) Getting the support they need, modeled after a successful intervention for patient groups. Manualization is crucial for successful wider implementation. Sessions 9 and 10 will provide booster sessions in which the interventionist will assess current challenges for the caregiver, provide review, and emphasize further coping skills training that might assist the caregiver in managing current stressors
Period: Overall Study
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Started | 83 | 76
Month 1.5 (Post Transplantation) | 79 | 76
Month 3 (Post Transplantation) | 66 | 62
Month 6 (Post Transplantation) | 63 | 52
Completed | 47 | 37
Not Completed | 36 | 39
Not completed — Withdrawal by Subject | 17 | 24
Not completed — Lost to Follow-up | 16 | 13
Not completed — Screen Failure | 3 | 1
Not completed — Patient did not receive transplant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0) | Total
Number analyzed (Participants) | 83 | 76 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Caregiver information was not available for TAU for the following variable: age (n = 2). PEPRR for the following variables: age (n = 1).
  years
    number analyzed (Participants) | 81 | 75 | 156
    (all) | 54.6 (12.8) | 53.6 (14.7) | 54.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Caregiver information was not available for TAU for the following variable: sex (n = 2). PEPRR for the following variables: sex (n = 1).
  Participants
    number analyzed (Participants) | 81 | 75 | 156
    Female | 67 | 58 | 125
    Male | 14 | 17 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 64 | 65 | 129
  Unknown or Not Reported | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 68 | 62 | 130
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 83 | 76 | 159
Annual income [Count of Participants; unit: Participants]
  < 25,000 | 29 | 21 | 50
  25,000-44,999 | 14 | 13 | 27
  45,000-64,999 | 13 | 18 | 31
  > 65,000 | 13 | 16 | 29
  Unknown or Not Reported | 14 | 8 | 22
Relationship to patient [Count of Participants; unit: Participants]
  Spouse/Civil Partner | 54 | 48 | 102
  Sibling | 5 | 8 | 13
  Parent | 11 | 9 | 20
  Child | 6 | 3 | 9
  Other | 0 | 7 | 7
  Unknown or Not Reported | 7 | 1 | 8
Employment Status (Before Caregiving) [Count of Participants; unit: Participants]
  Full-time | 30 | 35 | 65
  Part-time | 15 | 12 | 27
  Unemployed | 9 | 7 | 16
  On leave | 1 | 1 | 2
  Retired | 20 | 20 | 40
  Unknown or Not Reported | 8 | 1 | 9
Employment Status (During Caregiving) [Count of Participants; unit: Participants]
  Full-time | 15 | 18 | 33
  Part-time | 15 | 14 | 29
  Unemployed | 9 | 12 | 21
  On leave | 15 | 13 | 28
  Retired | 20 | 17 | 37
  Unknown or Not Reported | 9 | 2 | 11
Patient Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (14.2) | 51.9 (15.3) | 53.3 (14.8)
Patient Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 54 | 49 | 103
Patient Diagnosis [Count of Participants; unit: Participants] — Abbreviations: MDS, myelodysplastic syndrome; MPS, myeloproliferative syndrome; MM, multiple myeloma; SAA, severe aplastic anemia.
  Participants
    Leukemia | 53 | 44 | 97
    Lymphoma | 11 | 10 | 21
    MDS/MPS | 16 | 19 | 35
    Other (MM, SAA) | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Functional Assessment of Cancer Treatment - Blood/Marrow Transplant
Description: "Functional Assessment of Cancer Treatment - Blood/Marrow Transplant" (FACT-BMT) is used to assess the life quality of patients. The scale includes 5 subscales. The scores of each scale are summed to compute a total score. The scale range is 0-148. Higher score indicates better life quality.
Time Frame: Baseline (prior to transplant), 6 weeks, 3 months and 6 months after transplant
Population: Patient Control group missing responses (n = 14). Caregiver Intervention group: missing responses (n = 6).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 69 | 70
units on a scale
  Baseline | 97.7 [93.3 to 102.2] | 98.1 [93.6 to 102.5]
  Month 1.5 | 95.7 [90.4 to 100.9] | 95.8 [90.3 to 101.2]
  Month 3 | 101.5 [96.2 to 106.8] | 100.1 [94.5 to 105.8]
  Month 6 | 100.9 [94.5 to 107.3] | 101.8 [94.2 to 109.4]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = .96, Mixed Models Analysis

2. Primary Outcome: Caregiver Distress - Principal Component Analysis
Description: Caregiver Distress is a composite score is created from a principal component analysis (PCA). This PCA extracted the first principal component from summary variables of Center for Epidemiological Studies Depression Scale, Spielberger State and Trait Anxiety Inventory, and Perceived Stress Scale. The composite distress score has a mean of 0.0 and SD of 1.0, scale ranges from -2.06 - 3.73. Higher score indicates greater distress.
Time Frame: Baseline (prior to transplant), 6 weeks, 3 months and 6 months after transplant
Population: Caregiver Control group missing responses (n = 7). Caregiver Intervention group: missing responses (n = 3).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 76 | 73
units on a scale
  Baseline | -0.09 [-0.31 to 0.14] | 0.07 [-0.16 to 0.30]
  Month 1.5 | 0.02 [-0.22 to 0.26] | -0.06 [-0.31 to 0.19]
  Month 3 | 0.05 [-0.21 to 0.32] | 0.0 [-0.27 to 0.28]
  Month 6 | 0.14 [-0.11 to 0.39] | -0.2 [-0.47 to 0.07]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.007, Mixed Models Analysis

3. Secondary Outcome: Perceived Stress Scale
Description: The "Perceived Stress Scale" (PSS) measures the overall level of stress. This instrument contains 14 items accessing overall appraisals of stress in the past month. The total score range is 0-56. A higher score indicates greater stress.
Time Frame: Baseline (prior to transplant), 6 weeks, 3 months and 6 months after transplant
Population: Caregiver Control group missing responses (n = 7). Caregiver Intervention group: missing responses (n = 3).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 76 | 73
units on a scale
  Baseline | 24.2 [22.3 to 26.1] | 25.5 [23.5 to 27.4]
  Month 1.5 | 23.0 [21.2 to 24.8] | 22.9 [21.1 to 24.8]
  Month 3 | 21.3 [19.2 to 23.5] | 22.4 [20.1 to 24.6]
  Month 6 | 21.9 [19.9 to 24.0] | 20.5 [18.3 to 22.7]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.08, Mixed Models Analysis

4. Secondary Outcome: Center for Epidemiological Studies Depression Scale
Description: "Center for Epidemiological Studies Depression" Scale (CESD) is a self-report 20-item scale designed to measure current depressive symptoms. Total score range from 0-60, with a score at or above 16 reflecting significant depressive symptomatology.
Time Frame: Baseline (prior to transplant), 6 weeks, 3 months and 6 months after transplant
Population: Caregiver Control group missing responses (n = 7). Caregiver Intervention group: missing responses (n = 3).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 76 | 73
units on a scale
  Baseline | 20.0 [18.5 to 21.4] | 20.5 [19.0 to 22.0]
  Month 1.5 | 19.6 [18.3 to 21.0] | 18.3 [16.9 to 19.7]
  Month 3 | 20.0 [18.3 to 21.7] | 17.8 [16.0 to 19.7]
  Month 6 | 21.3 [19.4 to 23.2] | 18.0 [16.0 to 20.0]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.05, Mixed Models Analysis

5. Secondary Outcome: Spielberger State-Trait Anxiety Inventory
Description: The "Spielberger State and Trait Anxiety Inventory" (STAI) is a validated self-reporting instrument used to assess anxiety in adults. The inventory consists of state anxiety, which evaluates how the subject feels currently (transient anxiety). The scale consists of 20 questions, and a higher score indicates greater anxiety. Total score ranges from 20 (no anxiety) to 80 (maximum anxiety).
Time Frame: Baseline (prior to transplant), 6 weeks, 3 months and 6 months after transplant
Population: Caregiver Control group missing responses (n = 7). Caregiver Intervention group: missing responses (n = 3).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 76 | 73
units on a scale
  Baseline | 39.6 [36.7 to 42.5] | 41.6 [38.6 to 44.6]
  Month 1.5 | 38.4 [35.4 to 41.3] | 39.6 [36.5 to 42.6]
  Month 3 | 39.2 [35.9 to 42.6] | 39.3 [35.8 to 42.8]
  Month 6 | 39.1 [35.8 to 42.4] | 35.7 [32.2 to 39.2]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.070, Mixed Models Analysis

6. Secondary Outcome: Change in Adrenal Activity Over Time
Description: Cortisol measured in hair will be used as a retrospective measure of activation of the hypothalamic pituitary adrenal axis. Because hair cortisol were not normally distributed, the data were log transformed.
Time Frame: Baseline (prior to transplant), 3 months (caregiver only), and 6 months after transplant.
Population: Caregiver Control group missing responses (n = 8). Caregiver Intervention group: missing responses (n = 2).
Measure: Least Squares Mean (95% Confidence Interval); unit: log (pg/mg)
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 75 | 74
log (pg/mg)
  Baseline | 1.93 [1.68 to 2.20] | 2.14 [1.88 to 2.40]
  Month 3 | 1.98 [1.71 to 2.26] | 2.18 [1.89 to 2.46]
  Month 6 | 2.19 [1.89 to 2.50] | 2.14 [1.80 to 2.47]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.96, Mixed Models Analysis

7. Secondary Outcome: Change in Caregiver Telomere Length Over Time
Description: Telomere length was assessed as a measure of cellular aging in blood samples from participants. Because telomere length were not normally distributed, the data were log transformed.
Time Frame: Baseline (prior to transplant), 3 months and 6 months after transplant
Population: Caregiver Control group missing responses (n = 8). Caregiver Intervention group: missing responses (n = 2).
Measure: Least Squares Mean (95% Confidence Interval); unit: log (T/S ratio)
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 75 | 74
log (T/S ratio)
  Baseline | 0.03 [-0.02 to 0.08] | 0.0 [-0.05 to 0.05]
  Month 3 | 0.03 [-0.02 to 0.08] | 0.0 [-0.05 to 0.06]
  Month 6 | 0.03 [-0.02 to 0.09] | 0.03 [-0.03 to 0.09]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.74, Mixed Models Analysis

8. Secondary Outcome: Change in Caregiver Telomerase Activity Over Time
Description: Telomerase activity will be assessed as a measure of the ability to reverse cellular aging processes. Because telomerase activity were not normally distributed, the data were log transformed.
Time Frame: Baseline (prior to transplant), 3 months and 6 months after transplant
Population: Caregiver Control group missing responses (n = 8). Caregiver Intervention group: missing responses (n = 2).
Measure: Least Squares Mean (95% Confidence Interval); unit: log (enzyme unit)
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 75 | 74
log (enzyme unit)
  Baseline | 1.7 [1.55 to 1.84] | 1.7 [1.56 to 1.85]
  Month 3 | 1.69 [1.57 to 1.82] | 1.73 [1.60 to 1.87]
  Month 6 | 1.76 [1.55 to 1.97] | 1.71 [1.47 to 1.95]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.79, Mixed Models Analysis

9. Secondary Outcome: Caregiver Reaction Assessment
Description: The "Caregiver Reaction Assessment" (CRA) is a measure of caregiver burden. This instrument contains 24 items reflecting the total caregiver situation in the past month. The scale includes 5 subscales. The scores of each scale are summed to compute a total score. Minimum score (best value)=5. Maximum score (worst value)=25. Higher values reflect the experience of a higher burden.
Time Frame: Baseline (prior to transplant), 6 weeks, 3 months and 6 months after transplant
Population: Caregiver Control group missing responses (n = 7). Caregiver Intervention group: missing responses (n = 3).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
Number analyzed (Participants) | 76 | 73
units on a scale
  Baseline | 10.4 [9.9 to 11.0] | 10.3 [9.7 to 10.9]
  Month 1.5 | 10.8 [10.1 to 11.4] | 10.9 [10.3 to 11.6]
  Month 3 | 10.8 [10.0 to 11.5] | 10.9 [10.2 to 11.7]
  Month 6 | 10.5 [9.7 to 11.4] | 10.5 [9.6 to 11.3]
Statistical Analysis 1: Comparison: Caregiver Self-Directed (TAU) vs Caregiver Intervention (PEPRR 2.0); Test type: Superiority; p = 0.86, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 years, 3 months
Arm/Group | Caregiver Self-Directed (TAU) | Caregiver Intervention (PEPRR 2.0)
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/76
Other Adverse Events (participants affected / at risk) | 0/83 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT02037568/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT02037568/Prot_SAP_001.pdf